CLINICAL TRIAL: NCT03836066
Title: A Phase II Open Label Study of Atezolizumab in Combination With Bevacizumab as First Line Treatment for Locally Advanced or Metastasic High-intermediate Tumor Mutation Burden Selected Non-squamous Non-small Cell Lung Cancer Patients.
Brief Title: Atezolizumab Plus Bevacizumab in First Line NSCLC Patients
Acronym: TELMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 18/03_TELMA; 2018-004654-17 (EudraCT Number)
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC, Atezolizumab, Bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Atezolizumab plus Bevacizumab arm (Experimental): 1 group, Atezolizumab 1200mb + Bevacizumab 15 mg/kg (IV),every 21 days.
  Interventions: Drug: Atezolizumab-Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab-Bevacizumab — Atezoluzumab 1200 mg + Bevacizumab 15 mg / kg
  Other Names: Tecentriq-Avastin

SUMMARY:
This is a multi-center phase II clinical trial of atezolizumab in combination with bevacizumab as first line treatment for locally advanced or metastasic high-intermediate tumour mutation burden selected NSCLC patients. 102 patients will be enrolled in this trial to examine the efficacy of this combination measured by progression free survival according to response evaluation Criteria in solid tumours (RECIST) version 1.1.

DETAILED DESCRIPTION:
Chemotherapy-naïve patients high-intermediate TMB (TMB≥10 mutations/MB) and with locally advanced or metastatic non-squamous non-small cell lung cancer patients will be selected. Enroled patientswill receive 1200 mg of atezolizumab and 15mg/Kg of Avastin® (bevacizumab) administered by IV infusion every 21 days (+/- 3 days).

The treatment will start within 1-5 days from enrolment. Atezolizumab may continue beyond disease progression per RECIST v1.1 until loss of clinical benefit, unacceptable toxicity, patient or physician decision to discontinue , or death. Bevacizumab will be administered until progression disease, unacceptable toxicity, patient or physician decision to discontinue or death.

For all patients, tumour response data collection will continue until disease progression, even if the patient stops study treatment prior to disease progression.

The primary endpoint is to evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by Progression Free Survival according to RECIST Version 1.1.

PFS after enrolment is defined as the time from enrolment to the first occurrence of disease progression or death from any cause, whichever occurs first.

Patient accrual is expected to be completed within 1.5 years excluding a run-in-period of 46 months. Treatment and follow-up are expected to extend the study duration to a total of 4.5 years. Patients will be followed 1.5 years after the end of treatment independently of the cause of end of treatment. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years old
2. ECOG performance status of 0 or 1.
3. Histologically or cytologically confirmed, Stage IIIB or IV non-squamous NSCLC according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology
4. No prior treatment for Stage IIIB or IV non-squamous NSCLC.
5. Patients who have received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy, or chemo-radiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from randomization since the last chemotherapy, radiotherapy, or chemo-radiotherapy.
6. Patients with a treated asymptomatic CNS metastasis are eligible, provided they meet all of the following criteria:

   1. Only supratentorial and cerebellar metastases allowed (i.e., no metastases to midbrain, pons, medulla or spinal cord).
   2. No ongoing requirement for corticosteroids as therapy for CNS disease.
   3. No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to randomization.
   4. No evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study. Patients with new asymptomatic CNS metastases detected at the screening scan must receive radiation therapy and/or surgery for CNS metastases. Following treatment, these patients may then be eligible without the need for an additional brain scan prior to inclusion, if all other criteria are met.
7. Patients with high-intermediate Tumour Mutational Burden analysed by Foundation Medicine (≥10 mutations/ MB) performed by a Foundation Medicine laboratory on previously obtained archival tumour tissue or tissue obtained from a biopsy at prescreening (sample must fulfil minimal sample requirements of 20% tumour cellularity and a minimum surface of 25mm2).
8. Measurable disease, as defined by RECIST v1.1. Previously irradiated lesions can only be considered as measurable disease if disease progression has been unequivocally documented at that site since radiation and the previously irradiated lesion is not the only site of disease.
9. Adequate hematologic and organ function defined by the following laboratory results obtained within 14 days prior to randomization:

   Neutrophils ≥ 1500 cells/μL without granulocyte colony-stimulating factor support.
   * Lymphocyte count ≥ 500/μL.
   * Platelet count ≥ 100,000/μL without transfusion.
   * Haemoglobin ≥ 9.0 g/dL. Patients may be transfused to meet this criterion.
   * INR or aPTT ≤ 1.5 × upper limit of normal (ULN). This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
   * AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN, with the following exceptions: Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN. Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 × ULN.
   * Serum bilirubin ≤ 1.25 × ULN. Patients with known Gilbert disease who have serum bilirubin level ≤ 3 × ULN may be enrolled.
   * Serum creatinine ≤ 1.5 × ULN or creatinine clearance of ≥45ml/min (based on the Cockcroft Gault formula).
10. All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention.
11. For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 5 months after the last dose of Atezolizumab and/or 6 months after the last dose of Bevacizumab, whichever is later. Such methods include: combined (oestrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD): intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
12. For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate [< 1% per year] when used consistently and correctly, and to continue its use for 6 months after the last dose of Bevacizumab. Male patients should not donate sperm during this study and for at least 6 months after the last dose of Bevacizumab.
13. Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drugs. The same rules are valid for male patients involved in this clinical study if they have a partner of childbirth potential. Male patients must always use a condom.
14. Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of study drug.

Exclusion Criteria:

1. Patients with a sensitizing mutation in the epidermal growth factor receptor (EGFR) gene.
2. Patients with an anaplastic lymphoma kinase (ALK) fusion oncogene.
3. Patients with an STK-1 Ligand alteration.
4. Patients with MDM2 amplification.
5. Patients with ROS1 translocations.
6. Active or untreated CNS metastases as determined by CT or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments.
7. Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to randomization.
8. Leptomeningeal disease.
9. Uncontrolled tumour-related pain. Patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should be treated prior to initiation of study drug. Patients should be recovered from the effects of radiation. There is no required minimum recovery period. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for locoregional therapy, if appropriate, prior to initiation of study drug.
10. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX®) are allowed.
11. Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN).
12. Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous-cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Principal Investigator — Hospital Universitario Puerta de Hierro
Locations (25):
- Spain (25):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - ICO Badalona, Badalona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Consorcio Hospitalario Provincial de Castelló, Castelló, Castelló
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Complejo Hospitalario de Jaén, Jaén, Jaén
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital La Princesa, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitario Son Llàtzer, Palma de Mallorca, Mallorca
  - Hospital General Universitario de Málaga, Málaga, Málaga
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Complejo Hospitalario de Toledo, Toledo, Toledo
  - Hospital Universitari i Politécnic La Fe, Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital General de Valencia, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Provencio M, Ortega AL, Coves-Sarto J, Calvo V, Marse-Fabregat R, Domine M, Guirado M, Carcereny E, Fernandez N, Alvarez R, Blanco R, Leon-Mateos L, Sanchez-Torres JM, Sullivan IG, Cobo M, Sanchez-Hernandez A, Massuti B, Sierra-Rodero B, Martinez-Toledo C, Serna-Blasco R, Romero A, Cruz-Bermudez A. Atezolizumab Plus Bevacizumab as First-line Treatment for Patients With Metastatic Nonsquamous Non-Small Cell Lung Cancer With High Tumor Mutation Burden: A Nonrandomized Controlled Trial. JAMA Oncol. 2023 Mar 1;9(3):344-353. doi: 10.1001/jamaoncol.2022.5959. PMID 36520426
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: Atezolizumab plus Bevacizumab arm
Started | 41
Completed | 38
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 307 patients were assessmed for elegibility but 266 were excluded for different reasons:
  * TMB < 10 (n=149)
  * TMB cannot be determined (n= 13)
  * No tumor/invalid sample (n= 24)
  * Insuficient sample (n= 21)
  * Other reasons (n= 59)
Arm/Group | Experimental: Atezolizumab Plus Bevacizumab Arm
Number analyzed (Participants) | 38
Age, Continuous [Mean (Full Range); unit: years] | 64.5 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Smoking habit [Count of Participants; unit: Participants]
  Non-smoker (≤ 100 cigarettes/lifetime) | 2
  Former smoker (≥ 1 year without smoking) | 21
  Smoker | 15
ECOG at diagnosis [Count of Participants; unit: Participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability GRADES: ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  Participants
    0 | 16
    1 | 22

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Atezolizumab in Combination With Bevacizumab - PFS
Description: To evaluate the efficacy of Atezolizumab in combination with Bevacizumab as measured by Progression Free Survival according to Response Evaluation Criteria in Solid Tumours (RECIST).
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
Population: A total of 41 patients were enrolled in this study. However, at the time of diagnosis, only 38 patients were analyzed, as 3 patients were excluded from the outcome measure studies. For the safety analysis, all enrolled patients (41) were included.
Measure: Median (Full Range); unit: Months
Arm/Group | Experimental: Atezolizumab plus Bevacizumab arm
Number analyzed (Participants) | 38
Months | 11.3 [8.1 to 16.5]

ADVERSE EVENTS:
Time Frame: From the subject's written consent to participate in the study through 30 days after the final administration of the IMP, up to 5 years
Description: A total of 41 patients had received treatment and were included in the safety analysis.
Arm/Group | Experimental: Atezolizumab plus Bevacizumab arm
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 13/41
Other Adverse Events (participants affected / at risk) | 20/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Atezolizumab plus Bevacizumab arm (N=41)
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Respiratory infection (Infections and infestations) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Nephritis (Renal and urinary disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Acute diverticulitis (Infections and infestations) | 1 (1)
AAA - suspected contained rupture (Vascular disorders) | 1 (1)
Left leg thrombophlebitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Atezolizumab plus Bevacizumab arm (N=41)
Fatigue (General disorders) | 2 (2)
Acute diverticulitis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Acute rectitis (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Serum amylase increased (Investigations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Arterial thromboembolism (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (6)
AAA - suspected contained rupture (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No study limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03836066/Prot_SAP_000.pdf